CLINICAL TRIAL: NCT00223405
Title: Analysis of Clinical Wear Patterns of Tooth Enamel and Ceramic Restorations as a Function of Particle Size, Inter-Particle Spacing and Fracture Toughness of Ceramic Crystals
Brief Title: Analysis of Enamel Wear Against Ceramic Restorations
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Ivoclar Vivadent AG (Industry); University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 012-1901-369; 116163; NCT01128231 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2013-04

CONDITIONS: Tooth Wear
Keywords: enamel wear against ceramic crowns
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- metal-ceramic (D'Sign) o: Metal ceramic crown will be placed
  Interventions: Device: crown placement
- an all-ceramic crown (IPS Empress2, Eris EXC).: All ceramic crown will be placed
  Interventions: Device: crown placement

INTERVENTIONS:
Device: crown placement

SUMMARY:
1. To characterize the microstructure (fracture toughness, particle size of ceramic, and inter-particle spacing) of three ceramic materials
2. To test the hypothesis that lower fracture toughness of glass and/or crystal phase in ceramics reduce wear damage of enamel.
3. To test the hypothesis that smaller sized crystals reduce wear damage of enamel.
4. To test the hypothesis that larger inter-particle spacing reduces wear damage of enamel.
5. To test the hypothesis that equivalent wear patterns exist in all directions between enamel versus enamel and ceramic versus enamel.
6. To test the hypothesis that bite force does not correlate with wear rates.
7. To test the hypothesis that salivary flow does not correlate with wear rates.
8. To test the hypothesis that a greater amount of wear is not associated with a loss in vertical dimension of occlusion.
9. To test the hypothesis that a greater amount of wear does not correlate with secondary cementum deposition as part of the passive eruption process.
10. To test the hypothesis that maximum wear occurs early and wear rates level off within the first two years.
11. To test the hypothesis that in vitro wear analysis does not correlate with in vivo wear measurements

DETAILED DESCRIPTION:
A total of 36 teeth (1 crown per patient) needing crowns will be selected with the following acceptance criteria:

1. Subjects must be over 18 years of age with good overall health. No contraindications to dental treatment must be present.
2. Subjects must have overall good dental health with no active tooth decay (caries) present and no periodontal disease. Pocket depth on all remaining teeth must not be more than 4 mm.
3. Subjects must have no existing temporomandibular disorder, (e.g. clicking, popping, pain on opening) or parafunctional habits (e.g. bruxism, clenching)
4. Subjects must need a crown on either a second premolar, first molar or second molar on any arch. Abutment teeth must be restorable and have a crown root ratio of at least 1:1. Abutment teeth must have a complement of opposing non-restored or minimally restored natural teeth. Minimally restored means nothing beyond a Class II amalgam restoration. Opposing arch cannot be a full coverage restoration or a partial denture. Contralateral tooth must be preferably present.
5. Subjects must exhibit good oral hygiene and compliance.
6. Subjects must not have any existing condition that could limit the flow of saliva; e.g. saliva flow must be of normal quantity.

Baseline data will be collected and will consist of:

1. General medical history and physical examination
2. Primary casts taken with polyvinylsiloxane impression material
3. Bite force measurement in Newtons using a gnathodynamometer
4. Pocket depths of abutment teeth must be recorded
5. Periapical radiographs of abutment teeth. Radiographs will be taken at the exact position with the use of the longitudinal radiographic analysis (LRA) technique.
6. Vertical dimension measured from the nasion to the lowest point on the chin
7. A saliva sample will be collected to ascertain quality (viscosity) and quantity. The parameters for analysis will be salivary pH, buffer capacity, secretion (ml/min), protein (mg/ml), phosphate (mmol/l), Ca (mval/l), Na (mval/l), K (mval/l).

A total of 36 teeth will be randomly assigned to receive either a metal-ceramic (D'Sign) or an all-ceramic crown (IPS Empress2, Eris EXC). Randomization will be done through a random number table. Teeth will be prepared by two operators: Dr. Josephine Esquivel-Upshaw and Dr. William Rose both from the General Dentistry department. Provisional restorations will be made from Integrity (Dentsply, USA) and final impressions will be made with a polyvinylsiloxane material using the two-stage technique. Master casts will be mounted in centric relation.

A single unit crown will be made from either two types of an all-ceramic material or a metal-ceramic material and cemented with a dual cure resin cement. Adjustments will be made with a high-speed handpiece and a fine diamond bur. Prior to cementation, all adjusted surfaces must be polished or glazed. Occlusal surface thickness of the crowns will be measured at baseline.

Baseline examination will be performed one week after cementation to ensure that the patient is comfortable with the crown and no further adjustments are needed. A polyvinylsiloxane impression will be made of the maxillary and mandibular arches to record the cemented crown and its antagonist arch.

The post-cementation casts will be poured with a Type IV gypsum product to enable proper scanning. A 3D Laserscanner will be used to scan in the x, y and z planes of tooth/teeth casts made from natural teeth. The vertical dimension will be recorded as well as periapical radiographs taken of the abutment teeth.

The subjects will be asked to return after six months of cementation. Polyvinylsiloxane impressions will once again be made of maxillary and mandibular arches and poured with Type IV stone. The antagonist teeth and the crown will be scanned using the 3D Laserscanner. Superimposition of baseline image and the six-month image will be performed and the amount of wear in three dimensions calculated mathematically. Vertical dimension of occlusion will also be determined by measurement of nasion to the lowest point on the chin and periapical radiographs taken of the restored teeth using the LRA technique. This procedure will be repeated every year for the next four years.

The amount of wear in microns will be determined for the x, y and z axes. Data will be subjected to a one-way ANOVA (α = 0.05 ) to determine any significant difference in wear of natural antagonist teeth and the ceramic crowns between baseline and yearly 3D images and also differences in wear between the yearly 3D images. Occlusal thickness of restorations will be determined based on the amount of wear calculated. Any presence of cracks or fractures will be recorded. Correlation of the amount of wear and any changes in vertical dimension and root cementum length will also be determined by comparison of nasion-chin height at different intervals.

ELIGIBILITY:
Inclusion Criteria:

Subjects needing a crown on a posterior tooth that is opposed by a natural tooth.

Exclusion Criteria:

1. Subjects must be over 18 years of age with good overall health. No contraindications to dental treatment must be present.
2. Subjects must have overall good dental health with no active tooth decay (caries) present and no periodontal disease. Pocket depth on all remaining teeth must not be more than 4 mm.
3. Subjects must have no existing temporomandibular disorder, (e.g. clicking, popping, pain on opening) or parafunctional habits (e.g. bruxism, clenching)
4. Subjects must need a crown on either a second premolar, first molar or second molar on any arch. Abutment teeth must be restorable and have a crown root ratio of at least 1:1. Abutment teeth must have a complement of opposing non-restored or minimally restored natural teeth. Minimally restored means nothing beyond a Class II amalgam restoration. Opposing arch cannot be a full coverage restoration or a partial denture. Contralateral tooth must be preferably present.
5. Subjects must exhibit good oral hygiene and compliance.
6. Subjects must not have any existing condition that could limit the flow of saliva; e.g. saliva flow must be of normal quantity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients needing a crown on a tooth that was opposed by a natural tooth. Patients seeking care in the UTHSCSA dental clinic.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2003-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
wear of the opposing enamel will be measured yearly for four years | up to 4 years

SECONDARY OUTCOMES:
wear of ceramic in vivo | up to 4 years
improved function of crown | uo to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Esquivel-Upshaw, D.M.D.,M.S., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States